CLINICAL TRIAL: NCT04266795
Title: A Randomized, Open-label, Controlled, Phase 2 Study of Pevonedistat, Venetoclax, and Azacitidine Versus Venetoclax Plus Azacitidine in Adults With Newly Diagnosed Acute Myeloid Leukemia Who Are Unfit for Intensive Chemotherapy
Brief Title: A Study of Pevonedistat and Venetoclax Combined With Azacitidine to Treat Acute Myeloid Leukemia (AML) in Adults Unable to Receive Intensive Chemotherapy
Acronym: PEVENAZA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pevonedistat-2002; 2019-003117-33 (EudraCT Number); U1111-1239-7581 (Registry Identifier: WHO)
Record Dates: First submitted 2020-02-04; First posted 2020-02-12 (Actual); Results first posted 2023-09-18 (Actual); Last update posted 2025-10-21 (Actual); Status verified 2025-10

CONDITIONS: Acute Myeloid Leukemia (AML)
Keywords: Drug Therapy
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — pevonedistat; venetoclax; Azacitidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Venetoclax 100/200/400 mg + Azacitidine 75 mg/m^2 (Active Comparator): Venetoclax 100 mg tablet orally on Day 1; 200 mg on Day 2; thereafter, at 400 mg on Day 3 through Day 28 in Cycle 1 (cycle length= 28 days) and 400 mg on Days 1 through 28 in Cycle 2 and beyond if tolerated. Following the confirmation of remission in Cycle 1 or thereafter, venetoclax 400 mg was administered on Day 1 through 21 or 28 as per Investigator's discretion, plus azacitidine 75 mg/m^2 intravenous (IV) or subcutaneous (SC) dosing on Days 1 through 7 or Days 1 through 5, Days 8, and 9 in each cycle up to primary completion date: 06 September 2022.
  Interventions: Drug: Venetoclax; Drug: Azacitidine
- Pevonedistat 20 mg/m^2 + Venetoclax 100/200/400 mg + Azacitidine 75 mg/m^2 (Experimental): Pevonedistat 20 mg/m^2 as a 60-minute IV infusion on Days 1, 3, and 5 in each 28-day cycle plus venetoclax 100 mg tablet orally on Day 1; 200 mg on Day 2; thereafter, at 400 mg on Day 3 through Day 28 in Cycle 1 (cycle length= 28 days) and 400 mg on Days 1 through 28 in Cycle 2 and beyond if tolerated. Following the confirmation of remission in Cycle 1 or thereafter, venetoclax 400 mg was administered on Day 1 through 21 or 28 as per Investigator's discretion, plus azacitidine 75 mg/m^2 IV or SC dosing on Day 1 through 7 or Days 1 through 5, Days 8, and 9 in each cycle up to primary completion date: 06 September 2022.
  Interventions: Drug: Pevonedistat; Drug: Venetoclax; Drug: Azacitidine

INTERVENTIONS:
Drug: Pevonedistat — Pevonedistat IV infusion.
  Other Names: TAK-924; MLN4924
  Arms: Pevonedistat 20 mg/m^2 + Venetoclax 100/200/400 mg + Azacitidine 75 mg/m^2
Drug: Venetoclax — Venetoclax tablets.
Drug: Azacitidine — Azacitidine IV or SC injection.

SUMMARY:
The main aim is to see how the combination of pevonedistat + venetoclax + azacitidine compares to venetoclax + azacitidine in adults recently diagnosed with AML who are unable to be treated with intensive chemotherapy.

Participants will receive either pevonedistat + venetoclax + azacitidine or venetoclax + azacitidine in 28-day treatment cycles. Bone marrow samples (biopsy) will be collected throughout the study. Pevonedistat will be given as an intravenous (IV) infusion and Azacitidine will be given through IV or subcutaneous (under the skin).

Study treatments may continue as long as the participant is receiving benefit from it. Participants may choose to stop treatment at any time.

DETAILED DESCRIPTION:
The drug being tested in this study is called Pevonedistat. Pevonedistat is being tested to treat people who have AML. This study will compare the improvement in EFS in Arm A: Pevonedistat + Venetoclax + Azacitidine combination arm group when compared with Arm B: Venetoclax + Azacitidine.

The study will enroll approximately 164 patients. Participants will be randomly assigned in 1:1 ratio to one of the two treatment groups in 28-day treatment cycles and which will remain disclosed to the patient and study doctor during the study:

* Pevonedistat 20 mg/m^2 + Venetoclax 400 mg (ramp-up dose, Cycle 1 only: 100-400mg) + Azacitidine 75 mg/m^2
* Venetoclax 400 mg (ramp-up dose, Cycle 1 only: 100-400 mg) + Azacitidine 75 mg/m^2

This multi-center trial will be conducted worldwide. The overall time to participate in this study is approximately 3 years. Participants will attend the end-of-treatment visit 30 days after the last dose of study drug or before the start of subsequent anti-neoplastic therapy if that occurs sooner.

ELIGIBILITY:
Inclusion Criteria:

* Has morphologically confirmed diagnosis of AML (World Health Organization [WHO] criteria 2008). Participants may have newly diagnosed primary de novo AML or secondary AML (sAML), defined as AML after myelodysplastic syndromes (MDS) or myeloproliferative neoplasm (MPN), or therapy-related AML (t-AML) following cytotoxic therapy, and/or radiotherapy for a malignant or nonmalignant disease.
* Is unfit for treatment with a standard arabinosylcytosine (Ara-C) and anthracycline induction regimen due to age or co-morbidities defined by 1 of the following:

  * ≥75 years of age. OR
  * ≥18 to <75 years of age with at least one of the following:
* Eastern Cooperative Oncology Group (ECOG) performance status of 2 or 3.
* Severe cardiac disorder (e.g., congestive heart failure requiring treatment, ejection fraction ≤50%, or chronic stable angina).
* Severe pulmonary disorder (e.g., carbon monoxide lung diffusion capacity ≤65% or forced expiratory volume in 1 second ≤65%).
* Creatinine clearance (CrCl) <45 mL/min (but ≥30 mL/min as part of general eligibility criteria).
* Hepatic disorder with total bilirubin >1.5 times the upper limit of the normal range (ULN).
* Has clinical laboratory values within the following parameters (repeat within 3 days before the first dose of study drug if laboratory values used for randomization were obtained more than 3 days before the first dose of study drug):

  * Total bilirubin ≤1.5 times the ULN except in participants with Gilbert's syndrome. Participants with Gilbert's syndrome may enroll with direct bilirubin ≤3 times the ULN of the direct bilirubin. Elevated indirect bilirubin due to posttransfusion hemolysis is allowed.
  * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤3.0 times the ULN.
  * Creatinine clearance (CrCl) ≥30 mL/min (calculated by the Modification of Diet in Renal Disease [MDRD] Study equation).
  * Albumin >2.7 g/dL.
* White blood cell (WBC) count <25 × 10^9/L. Participants who are cytoreduced with leukapheresis or with hydroxyurea may be enrolled if they meet the eligibility criteria before starting therapy.

Exclusion Criteria:

* Has history of MPN with BCR-ABL1 translocation or AML with BCR-ABL1 translocation.
* Has genetic diagnosis of acute promyelocytic leukemia.
* Is eligible for intensive chemotherapy and/or allogeneic stem cell transplantation.
* Has extramedullary AML without evidence of bone marrow involvement.
* Had prior treatment with hypomethylating agents for AML (hypomethylating agent treatment for prior MDS is not exclusionary).
* Has clinical evidence of or history of central nervous system involvement by AML.
* Had diagnosed or treated for another malignancy (except for adequately treated carcinoma in situ of any organ or nonmelanoma skin cancer) within 1 year before randomization or previously diagnosed with another malignancy and have any evidence of residual disease that may compromise the administration of pevonedistat, venetoclax or azacitidine. Prior MDS is also allowed, but the participant cannot have received treatment for MDS within 14 days before first dose of any study drug.
* Has a WBC count ≥25 × 10^9/L
* Has uncontrolled human immunodeficiency virus (HIV) infection. Note: Known HIV positive participants who meet the following criteria will be considered eligible:

  * Cluster difference 4 (CD4) count >350 cells/mm^3.
  * Undetectable viral load.
  * Maintained on modern therapeutic regimens utilizing non-cytochrome P (CYP)-interactive agents.
  * No history of acquired immune deficiency syndrome (AIDS)-defining opportunistic infections.
* Participant is known to be positive for hepatitis B or C infection, with the exception of those with an undetectable viral load within 3 months (hepatitis B or C testing is not required for eligibility assessment).
* Has hepatic cirrhosis.
* Has uncontrolled coagulopathy or bleeding disorder.
* Has high blood pressure which cannot be controlled by standard treatments.
* Has prolonged rate QTc interval ≥500 msec, calculated according to institutional guidelines.
* Has left ventricular ejection fraction (LVEF) <40%, based on echocardiogram or multi gated acquisition (MUGA) scan at screening (data to be available within last 3 months of screening).
* As infection is a common feature of AML, participants with active infection are permitted to enroll provided that the infection is under control and no signs of systemic inflammatory response beyond low grade fever that makes participant clinically unstable in the opinion of the investigator. Participants with uncontrolled infection shall not be enrolled until infection is treated and brought under control.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 164 (Actual)
Dates: Start 2020-10-13 (Actual); Primary Completion 2022-09-06 (Actual); Study Completion 2025-10-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (57):
- United States (23):
  - Banner MD Anderson Cancer Center, Gilbert, Arizona
  - UC San Diego Moores Cancer Center, La Jolla, California
  - UC Irvine Medical Center, Orange, California
  - University of Miami Miller School of Medicine, Miami, Florida
  - AdventHealth (Florida Hospital) - Transplant Institute, Orlando, Florida
  - Norton Cancer Institute - Suburban, Louisville, Kentucky
  - Tulane Medical Center, New Orleans, Louisiana
  - Massachusetts General Hospital, Boston, Massachusetts
  - HCA Midwest Health - SCRI - PPDS, Kansas City, Missouri
  - Northwell Health Cancer Institute, Lake Success, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Stony Brook Medicine, Stony Brook, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - The University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Rhode Island Hospital, Providence, Rhode Island
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Houston Methodist Cancer Center, Houston, Texas
  - Joe Arrington Cancer Research and Treatment Center, Lubbock, Texas
  - Intermountain LDS Hospital, Salt Lake City, Utah
  - University of Virginia Health System, Charlottesville, Virginia
  - West Virginia University Hospital, Morgantown, West Virginia
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Canada (5):
  - University of Alberta, Edmonton, Alberta
  - Tom Baker Cancer Centre, Tom Baker Cancer Centre, Alberta
  - London Health Sciences Centre, London, Ontario
  - Ottawa Hospital, Ottawa, Ontario
  - Hopital de L'enfant Jesus, Québec, Quebec
- France (12):
  - Centre Hospitalier Le Mans, Le Mans, Sarthe
  - Hopital Avicenne, Bobigny
  - Institut dHematologie de Basse Normandie, Caen
  - CHU de Grenoble, Grenoble
  - CHRU Lille, Lille
  - CHRU Nantes, Nantes
  - CHU de Nice, Nice
  - Hopital Saint Antoine, Paris
  - Hopital Saint Louis, Paris
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - CHRU de Poitiers La Miletrie, Poitiers
  - EDOG - Institut Claudius Regaud - PPDS, Toulouse
- Italy (9):
  - Grande Ospedale Metropolitano Bianchi-Melacrino-Morelli, Reggio Calabria, Calabria
  - ASST di Monza - Azienda Ospedaliera San Gerardo, Monza, Lombardy
  - Istituto Clinico Humanitas, Rozzano, Milano
  - Azienda Sanitaria Ospedaliera S Luigi Gonzaga, Orbassano, Piedmont
  - Azienda Ospedaliera Citta della Salute e della Scienza di Torino, Turin, Piedmont
  - Ospedale Santa Maria Della Misericordia Di Perugia, Perugia, Umbria
  - Azienda Ospedaliero Universitaria Di Bologna - Policlinico S Orsola Malpighi, Bologna
  - Azienda Ospedaliera Universitaria Careggi, Florence
  - Fondazione IRCCS Policlinico San Matteo di Pavia, Pavia
- Poland (8):
  - Szpital Uniwersytecki w Krakowie, Krakow, Lesser Poland Voivodeship
  - MTZ Clinical Research Sp z o o, Warsaw, Masovian Voivodeship
  - Instytut Hematologii i Transfuzjologii, Warsaw, Masovian Voivodeship
  - Uniwersytecki Szpital Kliniczny w Bialymstoku, Bialystok, Podlaskie Voivodeship
  - Szpital Uniwersytecki Nr 2 im. Dr Jana Biziela w Bydgoszczy, Bydgoszcz
  - Uniwersyteckie Centrum Kliniczne, Gdansk
  - Samodzielny Publiczny Szpital Kliniczny nr 1 w Lublinie, Lublin
  - Wojewodzkie Wielospecjalistyczne Centrum Onkologii i Traumatologii im. M. Kopernika w Lodzi, Lodz, Łódź Voivodeship

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- [Derived] Short NJ, Wierzbowska A, Cluzeau T, Laribi K, Recher C, Czyz J, Ochrem B, Ades L, Gallego-Hernanz MP, Heiblig M, Audisio E, Zarzycka E, Li S, Ferenc N, Yeh T, Faller DV, Sedarati F, Papayannidis C. Azacitidine and venetoclax with or without pevonedistat in patients with newly diagnosed acute myeloid leukemia. Leuk Lymphoma. 2025 Mar;66(3):458-468. doi: 10.1080/10428194.2024.2431878. Epub 2024 Nov 28. PMID 39606906
- See also: To obtain more information about this study, click this link — https://clinicaltrials.takeda.com/study-detail/5f6b603d4db2bf003ab4a389?idFilter=%5B%22Pevonedistat-2002%22%5D

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 51 investigative sites in France, Italy, Poland, United States and Canada from 13 October 2020 to 05 January 2024. The data is reported for primary outcome measure up to primary completion date: 06 September 2022. This study is ongoing.
Pre-assignment Details: Participants with a diagnosis of Acute Myeloid Leukemia (AML) were randomized in a 1:1 ratio to receive either pevonedistat + venetoclax + azacytidine or venetoclax + azacitidine.
Period: Overall Study
Arm/Group | Venetoclax 100/200/400 mg + Azacitidine 75 mg/m^2 | Pevonedistat 20 mg/m^2 + Venetoclax 100/200/400 mg + Azacitidine 75 mg/m^2
Started | 81 | 83
Safety Population (Safety population was defined as all participants who received at least 1 dose of any of the study medications (pevonedistat, venetoclax, or azacitidine).) | 80 | 81
Completed | 0 | 0
Not Completed | 81 | 83
Not completed — Adverse Event | 10 | 19
Not completed — Death | 7 | 8
Not completed — Initiation of Hematopoietic Stem Cell Transplant | 6 | 2
Not completed — Protocol-Specified Withdrawal Criterion Met | 1 | 0
Not completed — Progressive Disease | 12 | 9
Not completed — Withdrawal by Patient | 5 | 6
Not completed — Disease Relapse | 3 | 6
Not completed — Reason not Specified | 12 | 10
Not completed — Participants Ongoing on Treatment | 25 | 23

BASELINE CHARACTERISTICS:
Population: Intent-to-Treat (ITT) population was defined as all participants who were randomized.
Groups:
- Venetoclax 100/200/400 mg + Azacitidine 75 mg/m^2: Venetoclax 100 mg tablet orally on Day 1; 200 mg on Day 2; thereafter, at 400 mg on Day 3 through Day 28 in Cycle 1 (cycle length= 28 days) and 400 mg on Days 1 through 28 in Cycle 2 and beyond if tolerated. Following the confirmation of remission in Cycle 1 or thereafter, venetoclax 400 mg was administered on Day 1 through 21 or 28 as per Investigator's discretion, plus azacitidine 75 mg/m^2 IV or SC dosing on Days 1 through 7 or Days 1 through 5, Days 8, and 9 in each cycle up to primary completion date: 06 September 2022.
- Total: Total of all reporting groups
Arm/Group | Venetoclax 100/200/400 mg + Azacitidine 75 mg/m^2 | Pevonedistat 20 mg/m^2 + Venetoclax 100/200/400 mg + Azacitidine 75 mg/m^2 | Total
Number analyzed (Participants) | 81 | 83 | 164
Age, Continuous [Mean (Standard Deviation); unit: years] | 74.1 (5.99) | 74.5 (5.01) | 74.3 (5.50)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45 | 53 | 98
  Male | 36 | 30 | 66
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 2 | 3
  White | 56 | 64 | 120
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 24 | 17 | 41
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 3 | 6
  Not Hispanic or Latino | 50 | 60 | 110
  Not reported | 25 | 14 | 39
  Unknown | 3 | 6 | 9
Region of Enrollment [Count of Participants; unit: Participants]
  France | 23 | 25 | 48
  Italy | 22 | 20 | 42
  Poland | 18 | 16 | 34
  United States | 14 | 14 | 28
  Canada | 4 | 8 | 12

OUTCOME MEASURES:

1. Primary Outcome: Event-Free Survival (EFS)
Description: EFS was defined as time from study randomization to date of failure to achieve complete remission (CR)/CR with incomplete blood count recovery (CRi), relapse from CR/CRi, or death. Assessments of disease response based on criteria: European Leukemia Net (ELN) 2017 guidelines. CR was defined as bone marrow blasts <5%; absence of circulating blasts and blasts with Auer rods; absence of extramedullary disease; absolute neutrophil count (ANC)≥1.0×10^9/L (1000/µL); platelet count≥100×10^9/L (100,000/µL). CRi was defined as all CR criteria except for residual neutropenia (<1.0×10^9/L [1000/µL]) or thrombocytopenia (<100×10^9/L [100,000/µL]). For participants who achieved CR/CRi, if relapse is not observed by time of analysis, was censored at the date of last disease assessment. If failed to achieve CR/CRi, date of treatment failure was set on day of randomization.
Time Frame: Up to 22 months
Population: ITT population was defined as all participants who were randomized.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Venetoclax 100/200/400 mg + Azacitidine 75 mg/m^2 | Pevonedistat 20 mg/m^2 + Venetoclax 100/200/400 mg + Azacitidine 75 mg/m^2
Number analyzed (Participants) | 81 | 83
months | 11.24 [5.75 to NA] — The upper limit of 95% confidence interval was not estimable due to insufficient number of participants with events. | 7.72 [5.65 to NA] — The upper limit of 95% confidence interval was not estimable due to insufficient number of participants with events.
Statistical Analysis 1: Comparison: Venetoclax 100/200/400 mg + Azacitidine 75 mg/m^2 vs Pevonedistat 20 mg/m^2 + Venetoclax 100/200/400 mg + Azacitidine 75 mg/m^2; Test type: Superiority; p = 0.477, Log Rank; P-value was comparison of EFS between treatment groups and was based on the 1-sided stratified log-rank test statistic; Hazard Ratio (HR) = 0.99, 95% CI 2-sided [0.61 to 1.60] — Hazard ratio was based on an unadjusted stratified Cox proportional hazard regression model with stratification factors (randomization strata of age and AML subtype) and treatment as a factor in the model

2. Secondary Outcome: Overall Survival (OS)
Description: OS is defined as time from randomization to death from any cause. Participants without documentation of death at the time of analysis will be censored at the date last known to be alive.
Time Frame: Up to 36 months
Reporting Status: Not Posted, anticipated posting 2026-06

3. Secondary Outcome: Thirty-day Mortality Rate
Description: Mortality rate is defined as percentage of participants who survive at most 30 days from the first dose of study drug.
Time Frame: Day 30
Reporting Status: Not Posted, anticipated posting 2026-06

4. Secondary Outcome: Sixty-day Mortality Rate
Description: Mortality rate is defined as percentage of participants who survive at most 60 days from the first dose of study drug.
Time Frame: Day 60
Reporting Status: Not Posted, anticipated posting 2026-06

5. Secondary Outcome: Percentage of Participants With Complete Remission (CR)
Description: CR rate is defined as the percentage of participants who achieve the CR as evaluated by the investigator. Assessments of disease response are based on the criteria outlined in the ELN 2017 guidelines. CR is defined as bone marrow blasts <5%; absence of circulating blasts and blasts with Auer rods; absence of extramedullary disease; ANC≥1.0×10^9/L (1000/µL); platelet count≥100×10^9/L (100,000/µL).
Time Frame: Up to 36 months
Reporting Status: Not Posted, anticipated posting 2026-06

6. Secondary Outcome: Percentage of Participants With Composite Complete Remission (CCR)
Description: CCR rate is defined as the percentage of participants who achieve the CR + CRi as evaluated by the investigator. Assessments of disease response are based on the criteria outlined in the ELN 2017 guidelines. CR is defined as bone marrow blasts <5%; absence of circulating blasts and blasts with Auer rods; absence of extramedullary disease; ANC≥1.0×10^9/L (1000/µL); platelet count≥100×10^9/L (100,000/µL). CRi is defined as all CR criteria except for residual neutropenia (<1.0×10^9/L [1000/µL]) or thrombocytopenia (<100×10^9/L [100,000/µL]).
Time Frame: Up to 36 months
Reporting Status: Not Posted, anticipated posting 2026-06

7. Secondary Outcome: Overall Response Rate (ORR)
Description: ORR is defined as the percentage of participants who achieve the CR + CRi + Partial Remission (PR) as evaluated by the investigator. Assessments of disease response are based on the criteria outlined in the ELN 2017 guidelines. CR is defined as bone marrow blasts <5%; absence of circulating blasts and blasts with Auer rods; absence of extramedullary disease; ANC≥1.0×10^9/L (1000/µL); platelet count≥100×10^9/L (100,000/µL). CRi is defined as all CR criteria except for residual neutropenia (<1.0×10^9/L [1000/µL]) or thrombocytopenia (<100×10^9/L [100,000/µL]). PR is defined as all hematologic criteria of CR; decrease of bone marrow blast percentage to 5% to 25%; and decrease of pretreatment bone marrow blast percentage by at least 50%.
Time Frame: Up to 36 months
Reporting Status: Not Posted, anticipated posting 2026-06

8. Secondary Outcome: Percentage of Participants With CR + CRh
Description: CR + CRh rate is defined as the percentage of participants who achieve the CR + CRh as evaluated by the investigator. Assessments of disease response are based on the criteria outlined in the ELN 2017 guidelines. CR is defined as bone marrow blasts <5%; absence of circulating blasts and blasts with Auer rods; absence of extramedullary disease; ANC≥1.0×10^9/L (1000/µL); platelet count≥100×10^9/L (100,000/µL). CRh is defined as bone marrow with <5% blasts, peripheral blood neutrophil count >0.5×10^3/µL and peripheral blood platelet count >0.5×10^5/µL.
Time Frame: Up to 36 months
Reporting Status: Not Posted, anticipated posting 2026-06

9. Secondary Outcome: Percentage of Participants With Leukemia Response
Description: Leukemia response rate is defined as the percentage of participants who achieve the CR + CRi + PR + morphological leukemia-free state [MLFS, marrow CR (mCR)]) as evaluated by the investigator. Assessments of disease response are based on the criteria outlined in the ELN 2017 guidelines. CR is defined as bone marrow blasts <5%; absence of circulating blasts and blasts with Auer rods; absence of extramedullary disease; ANC≥ 1.0×10^9/L (1000/µL); platelet count≥100×10^9/L (100,000/µL). CRi is defined as all CR criteria except for residual neutropenia (<1.0×10^9/L [1000/µL]) or thrombocytopenia (<100×10^9/L [100,000/µL]). PR is defined as all hematologic criteria of CR; decrease of bone marrow blast percentage to 5% to 25%; and decrease of pretreatment bone marrow blast percentage by at least 50%. MLFS is defined as bone marrow blasts <5%; absence of blasts with Auer rods; absence of extramedullary disease; no hematologic recovery required.
Time Frame: Up to 36 months
Reporting Status: Not Posted, anticipated posting 2026-06

10. Secondary Outcome: Duration of CR and CRi
Description: Duration of CR and CRi is defined as the time from first documentation of CR or CRi to the date of first documentation of PD or relapse from CR or CRi, and will be summarized descriptively using the K-M method based on the responders. Assessments of disease response are based on the criteria outlined in the ELN 2017 guidelines. CR is defined as bone marrow blasts <5%; absence of circulating blasts and blasts with Auer rods; absence of extramedullary disease; ANC≥ 1.0×10^9/L (1000/µL); platelet count≥100×10^9/L (100,000/µL). CRi is defined as all CR criteria except for residual neutropenia (<1.0×10^9/L [1000/µL]) or thrombocytopenia (<100×10^9/L [100,000/µL]).
Time Frame: Up to 36 months
Reporting Status: Not Posted, anticipated posting 2026-06

11. Secondary Outcome: Time to First CR, CRi and PR
Description: Time to first CR, CRi, and PR is defined as the time from randomization until the first documented CR, CRi or PR, whichever occurs first, and will be analyzed using the K-M method. Assessments of disease response are based on the criteria outlined in the ELN 2017 guidelines. CR is defined as bone marrow blasts <5%; absence of circulating blasts and blasts with Auer rods; absence of extramedullary disease; ANC≥ 1.0×10^9/L (1000/µL); platelet count≥100×10^9/L (100,000/µL). CRi is defined as all CR criteria except for residual neutropenia (<1.0×10^9/L [1000/µL]) or thrombocytopenia (<100×10^9/L [100,000/µL]). PR is defined as all hematologic criteria of CR; decrease of bone marrow blast percentage to 5% to 25%; and decrease of pretreatment bone marrow blast percentage by at least 50%.
Time Frame: Up to 36 months
Reporting Status: Not Posted, anticipated posting 2026-06

12. Secondary Outcome: Plasma Concentration of Pevonedistat
Time Frame: At multiple time points pre-dose and post-dose on Days 1, 3 and 5 in Cycle 1 and post-dose on Day 1 in Cycles 2 and 4 (cycle length= 28 days)
Reporting Status: Not Posted, anticipated posting 2026-06

ADVERSE EVENTS:
Time Frame: From signing of informed consent to 30 days post last dose, up to primary completion date: 06 September 2022 (up to 22 months 24 days)
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment. Safety population was defined as all participants who received at least 1 dose of pevonedistat combination or azacitidine + venetoclax.
Arm/Group | Venetoclax 100/200/400 mg + Azacitidine 75 mg/m^2 | Pevonedistat 20 mg/m^2 + Venetoclax 100/200/400 mg + Azacitidine 75 mg/m^2
All-Cause Mortality (participants affected / at risk) | 15/80 | 18/81
Serious Adverse Events (participants affected / at risk) | 55/80 | 62/81
Other Adverse Events (participants affected / at risk) | 79/80 | 79/81
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Venetoclax 100/200/400 mg + Azacitidine 75 mg/m^2 (N=80) | Pevonedistat 20 mg/m^2 + Venetoclax 100/200/400 mg + Azacitidine 75 mg/m^2 (N=81)
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Acinetobacter bacteraemia (Infections and infestations) | 0 | 1
Acute coronary syndrome (Cardiac disorders) | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 4 | 1
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Acute myeloid leukaemia recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Altered state of consciousness (Nervous system disorders) | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 5 | 5
Arthritis bacterial (Infections and infestations) | 0 | 1
Asthenia (General disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0
Bacteraemia (Infections and infestations) | 1 | 1
Bacterial sepsis (Infections and infestations) | 0 | 1
Bradycardia (Cardiac disorders) | 1 | 0
Bronchitis bacterial (Infections and infestations) | 0 | 1
Bronchopulmonary aspergillosis (Infections and infestations) | 0 | 1
COVID-19 (Infections and infestations) | 2 | 2
COVID-19 pneumonia (Infections and infestations) | 1 | 1
Capillary leak syndrome (Vascular disorders) | 0 | 1
Cardiac arrest (Cardiac disorders) | 1 | 0
Cardiac failure (Cardiac disorders) | 0 | 3
Cardiac failure acute (Cardiac disorders) | 0 | 1
Cardiogenic shock (Cardiac disorders) | 0 | 1
Catheter site cellulitis (Infections and infestations) | 1 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 2
Clostridium difficile colitis (Infections and infestations) | 0 | 1
Clostridium difficile infection (Infections and infestations) | 0 | 1
Condition aggravated (General disorders) | 1 | 1
Cryptococcosis (Infections and infestations) | 1 | 0
Deafness neurosensory (Ear and labyrinth disorders) | 0 | 1
Death (General disorders) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Device related sepsis (Infections and infestations) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Diverticulitis (Infections and infestations) | 2 | 0
Enterobacter bacteraemia (Infections and infestations) | 0 | 1
Enterococcal bacteraemia (Infections and infestations) | 1 | 1
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 | 1
Escherichia bacteraemia (Infections and infestations) | 0 | 2
Escherichia sepsis (Infections and infestations) | 1 | 0
Failure to thrive (Metabolism and nutrition disorders) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 2 | 0
Fatigue (General disorders) | 0 | 1
Febrile bone marrow aplasia (Blood and lymphatic system disorders) | 2 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 20 | 14
Femur fracture (Injury, poisoning and procedural complications) | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
General physical health deterioration (General disorders) | 3 | 1
Haematoma (Vascular disorders) | 0 | 1
Haemorrhage intracranial (Nervous system disorders) | 1 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 1
Hyperleukocytosis (Blood and lymphatic system disorders) | 1 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1
Hypotension (Vascular disorders) | 1 | 1
Hypotensive crisis (Vascular disorders) | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Infection (Infections and infestations) | 0 | 1
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 0 | 1
Intervertebral discitis (Infections and infestations) | 1 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 1
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0
Metabolic acidosis (Metabolism and nutrition disorders) | 0 | 1
Multiple organ dysfunction syndrome (General disorders) | 2 | 2
Myelosuppression (Blood and lymphatic system disorders) | 0 | 1
Myocarditis (Cardiac disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 2
Neutropenic sepsis (Infections and infestations) | 2 | 1
Non-cardiac chest pain (General disorders) | 0 | 1
Pancytopenia (Blood and lymphatic system disorders) | 2 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 1
Platelet count decreased (Investigations) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonia (Infections and infestations) | 10 | 7
Pneumonia bacterial (Infections and infestations) | 1 | 0
Pneumonia fungal (Infections and infestations) | 1 | 1
Pneumonia legionella (Infections and infestations) | 1 | 0
Portal vein cavernous transformation (Hepatobiliary disorders) | 1 | 0
Proctalgia (Gastrointestinal disorders) | 1 | 0
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pyrexia (General disorders) | 4 | 5
Renal failure (Renal and urinary disorders) | 0 | 1
Respiratory acidosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory syncytial virus infection (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 7 | 6
Septic shock (Infections and infestations) | 2 | 5
Soft tissue inflammation (General disorders) | 1 | 0
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Staphylococcal bacteraemia (Infections and infestations) | 1 | 1
Subarachnoid haemorrhage (Nervous system disorders) | 0 | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 1 | 1
Syncope (Nervous system disorders) | 3 | 2
Systemic candida (Infections and infestations) | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 8 | 2
Toxic encephalopathy (Nervous system disorders) | 0 | 1
Tumour lysis syndrome (Metabolism and nutrition disorders) | 0 | 2
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Urinary retention (Renal and urinary disorders) | 1 | 0
Urinary tract infection (Infections and infestations) | 2 | 2
Vomiting (Gastrointestinal disorders) | 1 | 1
White blood cell count decreased (Investigations) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Venetoclax 100/200/400 mg + Azacitidine 75 mg/m^2 (N=80) | Pevonedistat 20 mg/m^2 + Venetoclax 100/200/400 mg + Azacitidine 75 mg/m^2 (N=81)
Abdominal pain (Gastrointestinal disorders) | 10 | 10
Alanine aminotransferase increased (Investigations) | 4 | 6
Anaemia (Blood and lymphatic system disorders) | 32 | 30
Anxiety (Psychiatric disorders) | 1 | 6
Arthralgia (Musculoskeletal and connective tissue disorders) | 8 | 10
Aspartate aminotransferase increased (Investigations) | 4 | 8
Asthenia (General disorders) | 16 | 14
Atrial fibrillation (Cardiac disorders) | 7 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 8 | 6
Blood bilirubin increased (Investigations) | 3 | 7
Blood creatinine increased (Investigations) | 12 | 8
Chills (General disorders) | 4 | 7
Constipation (Gastrointestinal disorders) | 26 | 34
Contusion (Injury, poisoning and procedural complications) | 5 | 6
Cough (Respiratory, thoracic and mediastinal disorders) | 7 | 5
Decreased appetite (Metabolism and nutrition disorders) | 15 | 8
Diarrhoea (Gastrointestinal disorders) | 25 | 28
Dizziness (Nervous system disorders) | 6 | 5
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 7 | 14
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 8 | 6
Fall (Injury, poisoning and procedural complications) | 2 | 6
Fatigue (General disorders) | 8 | 10
Febrile neutropenia (Blood and lymphatic system disorders) | 16 | 12
Haemorrhoids (Gastrointestinal disorders) | 9 | 6
Headache (Nervous system disorders) | 7 | 11
Hyperbilirubinaemia (Hepatobiliary disorders) | 4 | 6
Hyperkalaemia (Metabolism and nutrition disorders) | 7 | 8
Hyperphosphataemia (Metabolism and nutrition disorders) | 5 | 3
Hypertension (Vascular disorders) | 4 | 7
Hypoalbuminaemia (Metabolism and nutrition disorders) | 5 | 8
Hypocalcaemia (Metabolism and nutrition disorders) | 11 | 11
Hypokalaemia (Metabolism and nutrition disorders) | 26 | 26
Hypomagnesaemia (Metabolism and nutrition disorders) | 9 | 8
Hyponatraemia (Metabolism and nutrition disorders) | 6 | 9
Hypophosphataemia (Metabolism and nutrition disorders) | 6 | 12
Hypotension (Vascular disorders) | 10 | 12
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3 | 5
Injection site erythema (General disorders) | 6 | 2
Injection site pain (General disorders) | 5 | 2
Insomnia (Psychiatric disorders) | 8 | 6
Leukopenia (Blood and lymphatic system disorders) | 12 | 10
Lymphocyte count decreased (Investigations) | 5 | 4
Nausea (Gastrointestinal disorders) | 32 | 25
Neutropenia (Blood and lymphatic system disorders) | 46 | 47
Neutrophil count decreased (Investigations) | 8 | 7
Oedema peripheral (General disorders) | 12 | 18
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6 | 4
Platelet count decreased (Investigations) | 8 | 5
Pneumonia (Infections and infestations) | 7 | 12
Pruritus (Skin and subcutaneous tissue disorders) | 4 | 7
Pyrexia (General disorders) | 14 | 22
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 | 5
Thrombocytopenia (Blood and lymphatic system disorders) | 31 | 37
Tumour lysis syndrome (Metabolism and nutrition disorders) | 6 | 2
Vomiting (Gastrointestinal disorders) | 25 | 13
White blood cell count decreased (Investigations) | 7 | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.

DOCUMENTS (2):
  • Study Protocol (2022-01-21): https://cdn.clinicaltrials.gov/large-docs/95/NCT04266795/Prot_000.pdf
  • Statistical Analysis Plan (2022-06-22): https://cdn.clinicaltrials.gov/large-docs/95/NCT04266795/SAP_001.pdf